CLINICAL TRIAL: NCT05002881
Title: A Randomized, Double-blind, Cross-over, Placebo Controlled Study to Explore the Effect of Moringa Oleifera (E-HS-01) on Flow Mediated Dilatation and Hemodynamics
Brief Title: A Study to Explore the Effect of Moringa Oleifera (E-HS-01) on Flow Mediated Dilatation and Hemodynamics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: EB/210502/MO/FMD
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-10

CONDITIONS: Endothelial Function

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Cross-over, Placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, Cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa oleifera (E-HS-01) (Active Comparator): One capsule to be taken stat
  Interventions: Other: Moringa oleifera (E-HS-01); Other: Placebo
- Placebo (Placebo Comparator): One capsule to be taken stat
  Interventions: Other: Moringa oleifera (E-HS-01); Other: Placebo

INTERVENTIONS:
Other: Moringa oleifera (E-HS-01) — One capsule to be taken stat
Other: Placebo — One capsule to be taken stat

SUMMARY:
The present study is designed to evaluate the modulatory effect of IP on the vascular endothelial function. To assess its vasodilatation potential, change in flow mediated dilation (FMD) and blood flow velocity (BFV) will be assessed in healthy adult male population.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, physically active male volunteers aged between 20 to 35 years.
2. Body mass index (BMI) ≥ 20 and ≤ 29.9 kg/m2.
3. Participants with low to moderate physical activity as defined by a six-point scale score of ≥1 to ≤ 4.
4. Participants with systolic blood pressure (SBP) ≤ 139 and diastolic blood pressure (DBP) ≤ 89 mm Hg.
5. Ability to read and provide written, personally signed, and dated informed consent to participate in the study.
6. Ready to abstain from alcohol, caffeine, and vigorous physical activity (as assessed by six point scale) for 24 hours prior to every study visit.
7. Ready to abstain from beet root, moringa, and spinach for 48 hours prior to every study visit.

Exclusion Criteria:

1. Participants with history of pulmonary disorders (asthma, chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, pneumonia, etc)
2. Participants having fasting blood glucose (FBG) levels ≥ 125 mg/dL.
3. Participants currently on/or having history of taking antihypertensives / diuretics.
4. Smokers and tobacco users.
5. Participants with heavy alcohol consumption, defined as more than 14 standard alcoholic drink (SAD)/week or more than 4 SAD in a day.

   (NOTE - A standard alcoholic drink contains approximately 14 grams of alcohol, which is equivalent to 12 ounces of beer (~5% alcohol), 8.5 ounces of malt liquor (~9% alcohol), 5 ounces of wine (~12% alcohol), 3.5 ounces of fortified wine (e.g., sherry or port), or 1.5 ounces of liquor (distilled spirits; ~40% alcohol).
6. Participants currently on performance enhancing supplements.
7. History/symptoms of coronary artery disease, myocardial infarction etc.
8. Participants with any other condition which in the view of the investigator is likely to interfere with the study or put the participants at risk.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Percent flow mediated dilatation | From baseline (pre-IP administration) to 3 hours post-IP administration
  To determine change in the endothelial function after single dose administration of Moringa oleifera as assessed by the change in the Percent flow mediated dilatation of brachial artery, from baseline (pre-IP administration) to 3 hours post IP administration, in comparison to the placebo.

SECONDARY OUTCOMES:
Blood flow velocity | at baseline (pre-IP administration) and at 1, 2, and 3 hours post-IP administration
  The endothelial function can be assessed by measuring changes in blood flow by intravascular ultrasound. It has been demonstrated that biophysical forces such as flow-derived forces, modulates the vascular structure and function. Endothelium is mechanotransducer, which senses mechanical forces on its surface and the transduces these signals into biochemical signals. There exists a large body of literature regarding the wide spectra of biological signals induced by blood flow in the endothelium.18 Thus to evaluate the effect of Moringa oleifera on hemodynamics, change in blood flow velocity (cm/seconds) will be assessed at baseline (pre-IP administration) and at 1, 2, and 3 hours post-IP administration will be measured.
Percent flow mediated dilatation | at 1, and 2 hours post-IP administration from baseline (pre-IP administration)
  To identify the onset of effect of the investigational product, the flow mediated dilation at 1, and 2 hours post-IP administration from baseline (pre-IP administration) will be assessed as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dr, Anjali Jain, BHMS, Principal Investigator — Vedic lifesciences
Locations (1):
- Vedic Lifesciences, Mumbai, Maharashtra, India